CLINICAL TRIAL: NCT06724159
Title: PRINCIS Study ("Public Health Clinical Research Project"): Observational Study of the Effectiveness of Drugs Funded by the National Health System for Genitourinary Tumors.
Brief Title: Observational Study of the Effectiveness of Funded Drugs for Genitourinary Tumors.
Acronym: SOGUG-PRINCIS
Status: Recruiting | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: MFAR (Other)
Responsible Party: Sponsor
Other Study IDs: SOGUG-PRINCIS
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Genitourinary Cancers
Keywords: Urothelial carcinoma; Prostate adenocarcinoma; Renal carcinoma; Darolutamida; Nivolumab; Enfortumab Vedotin
MeSH Terms: conditions — Urogenital Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Renal Cell | interventions — darolutamide; enfortumab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TRIDA Cohort: Patients with hormone-sensitive prostate carcinoma not castrated who have started treatment with darolutamide in combination with androgen deprivation therapy and docetaxel, from January 1, 2024
  Interventions: Drug: darolutamide
- NIADY Cohort: Patients with urothelial carcinoma who have started treatment with adjuvant Nivolumab on or after August 1, 2023
  Interventions: Drug: Nivolumab monotherapy
- EV3aL Cohort: Patients with urothelial carcinoma who have started treatment with Enfortumab Vedotin (EV) on or after January 1, 2024
  Interventions: Drug: enfortumab vedotin

INTERVENTIONS:
Drug: darolutamide — Darolutamide in combination with androgen deprivation therapy and docetaxel. Following the posology and administration details of its marketing authorization and standard clinical practice
  Groups: TRIDA Cohort
Drug: Nivolumab monotherapy — Adjuvant nivolumab following after surgical removal of urothelial carcinoma. Following the posology and administration details of its marketing authorization and standard clinical practice
  Groups: NIADY Cohort
Drug: enfortumab vedotin — Following the posology and administration details of its marketing authorization and standard clinical practice
  Groups: EV3aL Cohort

SUMMARY:
SOGUG-PRINCIS is a retrospective (regarding patient inclusion) and prospective follow-up, epidemiological, non-interventional, non-blinded, non-randomized, multicenter, national observational study with drugs. This study will collect data from patients with genitourinary tumors to analyze the effectiveness under routine clinical practice conditions of drugs recently approved for funding in the Spanish National Health System.

In all cases, the decision to start treatment will be made prior to and independently of participation in the study, which will be limited to subsequently collecting the data necessary to assess the objectives of the study.

This study will serve as a registry for genitourinary cancers. Every time a new drug will be authorized, a new subproject with a primary endpoint will be opened to recruitment. The substudy will try to validate with real-world data the endpoints reported in the phase III clinical trials that led to the marketin authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Patients granting the ICF unless exemption or exceptions mentioned below.
* Histological diagnosis of malignant neoplasia originating in the genitourinary system: kidney, renal pelvis, ureter, bladder, prostate, testicle and germinal tissue of other locations, urethra, penis, or seminal vesicles.
* Patients have started treatment with medications whose positive resolution of financing by the Spanish National Health System for the aforementioned tumors has been after January 1, 2023.
* Patients have started treatment after the official publication of the positive resolution of financing of the drug under study by the National Health System. This restriction is intended to avoid interference of the study with the marketing authorization processes by the European Medicines Agency, and price and reimbursement negotiations by the Spanish health authorities.
* Patients have received treatment at the participating center.

Exclusion Criteria:

* Patients previously treated at another centre who have subsequently been referred to one of the participating centres. In this case, the patient will be included in the centre where treatment was started, or in the second centre if the first is not part of this study.
* Patients who do not meet any of the inclusion criteria.
* Evidence of an express objection by the subject or his/her legal representative to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with genitourinary cancers treated with new therapies following the standard clinical practice
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progresion-free survival rate at 18 months | 18 months after the initiation of study treatment
  For TRIDA substudy. Defined as the percentage of patients alive and free of progression of the disease (estimated by Kaplan-Meier method) at 18 months. Patients without event are censored in their last follow-up
Relapse-free survival rate at 24 months | 24 months after the first dose of study treatment
  For NIADY substudy. Defined as the percentage of patients alive and with no disease recurrence (estimated by Kaplan-Meier method) at 24 months
Overall survival rate at 12 months | 12 months after the first dose of study treatment
  For EV3aL substudy Defined as the percentage of patients alive (estimated by Kaplan-Meier method) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: José Ángel Arranz Arija, M.D.; Ph.D., Study Chair — Hospital General Universitario Gregorio Marañón de Madrid; Aránzazu González del Alba, M.D.; Ph.D., Study Chair — Hospital Universitario Puerta de Hierro; Sergio Vázquez Estévez, M.D.; Ph.D., Study Chair — Hospital Universitario Lucus Augusti
Locations (84):
- Spain (84):
  - Complejo Hospitalario Universitario de Albacete, Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Universitario Torrecárdenas, Almería, Andalusia
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Clínico San Cecilio, Granada, Andalusia
  - Hospital Universitario Virgen a de las Nieves, Granada, Andalusia
  - Hospital Universitario de Jaén, Jaén, Andalusia
  - Hospital Universitario Jerez de la Frontera, Jerez de la Frontera, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Quirón Salud Sagrado Corazón de Sevilla, Seville, Andalusia
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitario Virgen de Valme, Seville, Andalusia
  - Hospital Universitario San Jorge, Huesca, Aragon
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital General Mateu Orfila, Maó, Balearic Islands
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Cruces, Barakaldo, Basque Country
  - Hospital Universitario Basurto, Bilbao, Basque Country
  - OSI Donostialdea - Onkologikoa, Donostia / San Sebastian, Basque Country
  - Hospital Galdakao-Usansolo Ospitalea, Galdakao, Basque Country
  - Hospital Universitario de Álava - Txagorritxu, Vitoria-Gasteiz, Basque Country
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario de Burgos, Burgos, Castille and León
  - Complejo Hospitalario de Palencia, Palencia, Castille and León
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Castille and León
  - Hospital General de Segovia, Segovia, Castille and León
  - Hospital Clínico Universitario de Valladolid (HCUV), Valladolid, Castille and León
  - Complejo Hospitalario Zamora, Zamora, Castille and León
  - Hospital Universitario Mancha Centro, Alcázar de San Juan, Castille-La Mancha
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital Virgen de la Luz, Cuenca, Castille-La Mancha
  - Hospital Universitario de Guadalajara, Guadalajara, Castille-La Mancha
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall d'Hebrón, Barcelona, Catalonia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Catalonia
  - Hospital Universitari Parc Taulí, Sabadell, Sabadell, Catalonia
  - Hospital Universitari General de Catalunya, Sant Cugat Del Vallés, Catalonia
  - Hospital Universitario de Badajoz, Badajoz, Extremadura
  - Hospital San Pedro de Alcántara, Cáceres, Extremadura
  - Hospital Universitario de A Coruña (CHUAC), A Coruña, Galicia
  - Centro Oncológico de Galicia, A Coruña, Galicia
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Clínico Universitario de Santiago ~ CHUS, Santiago de Compostela, Galicia
  - Hospital Álvaro Cunqueiro, Vigo, Galicia
  - Hospital Universitario San Pedro, Logroño, La Rioja
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Central de la Defensa Gómez Ulla, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián, Madrid
  - Hospital Universitario Infanta Leonor, Vallecas, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Virgen de los Lirios, Alcoy, Valencia
  - Hospital Universitario de la Ribera, Alzira, Valencia
  - Hospital Universitario del Vinalopó, Elche, Valencia
  - Hospital General de Requena, Requena, Valencia
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario de Torrevieja, Torrevieja, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Consorcio Hospital General Universitario de València, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Marina Baixa, Villajoyosa, Valencia
  - Hospital Lluis Alcanyís de Xàtiva, Xàtiva, Valencia
  - Hospital Universitario de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
No IDP sharing is prestablished